CLINICAL TRIAL: NCT02526615
Title: Comparison of Effects of Rosiglitazone and Metformin on Myocardial, Skeletal Muscle, Liver and Adipose Tissue Insulin Stimulated Glucose Uptake in Patients With Type 2 Diabetes Mellitus
Brief Title: Effects of Rosiglitazone and Metformin on Metabolism in Type 2 Diabetes
Acronym: ROSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: SmithKline Beecham (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TurkuUH-ROSI
Record Dates: First submitted 2015-08-11; First posted 2015-08-18 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Insulin Sensitivity; Type 2 Diabetes
Keywords: rosiglitazone; metformin; muscle
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): placebo, 2 tablets per day
  Interventions: Drug: Placebo
- Metformin (Active Comparator): 500mg 1 tablet 2 times per day for the first 2 weeks, then after that 2 tables 2 times per day
  Interventions: Drug: Metformin
- Rosiglitazone (Active Comparator): 2 mg 1 tablets 2 times per day for the first 2 weeks, then after that 2 tablets 2 times per day
  Interventions: Drug: Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone — Patients received either placebo, metformin or rosiglitazone
  Other Names: Avandia
  Arms: Rosiglitazone
Drug: Metformin — Patients received either placebo, metformin or rosiglitazone
  Arms: Metformin
Drug: Placebo — Patients received either placebo, metformin or rosiglitazone
  Arms: Placebo

SUMMARY:
The objectives of this study are to compare the effects of rosiglitazone and metformin on insulin stimulated glucose uptake in subjects with type 2 diabetes. Whole body, and skeletal muscle, heart and adipose tissue insulin stimulated glucose uptake is measured during euglycemic hyperinsulinemic clamp and positron-emission tomography scanning before and 26 weeks after treatment in 48 newly diagnosed subjects with type 2 diabetes. Subjects will be randomized to receive either rosiglitazone or metformin or placebo, according to a simple randomization procedure with double blinding.

DETAILED DESCRIPTION:
Insulin resistance is a pivotal underlying metabolic abnormality in most subjects with type 2 diabetes. Clinical experience has proved metformin to be efficacious treatment in patients with type 2 diabetes. Rosiglitazone is a novel antidiabetic agent, which has been shown to decrease fasting plasma glucose concentrations in animal models and in clinical trials. There are no previous studies that compare the effects of rosiglitazone and metformin on insulin stimulated glucose uptake in subjects with type 2 diabetic in different organs.

PET is very sensitive in detecting changes in glucose uptake and blood flow and, is the method of choice to investigate the effects of medical interventions. Due to sensitivity of these functional parameters only moderate or small number of subjects need to be studied. This makes it feasible to perform tightly controlled intervention studies in a very cost-effective way.

The objectives of this study are to compare the effects of rosiglitazone and metformin on insulin stimulated glucose uptake in subjects with type 2 diabetes. PET measurements on myocardium, skeletal muscle and subcutaneous and visceral fat are performed at baseline and at the end of the treatment period. Furthermore, the effect of exercise on skeletal muscle blood flow and glucose uptake is studied.

The study consists of 48 newly diagnosed subjects with type 2 diabetes. Subjects will be randomized to receive either rosiglitazone or metformin or placebo, according to a simple randomization procedure with double blinding. The investigators will also study ten age-matched non-diabetic control subjects, who will undergo the same PET study procedure as subjects with type 2 diabetes.

A study of the effects of antidiabetic oral medication in newly diagnosed subjects with type 2 diabetes is of great importance for the understanding of the differences in mode of action of the different antidiabetic drugs. Such a study would contribute to elucidate advantages and disadvantages with certain drugs and potential additive effects in combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75 years,
* BMI 25-35 kg/m2,
* WHO criteria for type 2 diabetes fasting plasma glucose>=7.0 mmol/l on at least 2 separate occasions,
* C-peptide>0.2 nmol/l

Exclusion Criteria:

* plasma glucose < 6.1 or >10 mmol/l after the screening period
* cardiac heart failure
* diagnosed coronary heart disease
* severe aortic, mitral or tricuspidal valve disease
* blood pressure > 160/ 100 mg Hg
* any previous or present hepatic (GT >100, alanine amino transferase >3 x upper limit of the reference range) or renal (S-creatinine > 130) disease
* pregnancy or lactation
* proliferative retinopathy
* microalbuminuria
* subjects with history of lactate acidosis
* symptomatic polyneuropathy
* antidiabetic medication
* changes in antihypertensive medication or beta-blockers in medication
* metal objects in region of imaging
* anemia with Hb < 100 in mean or < 90 in women
* oral corticosteroid treatment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2000-10; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity in skeletal muscle | 26 weeks
  pre and at 26 weeks measured with euglycemic clamp and 18-F-2-fluoro-2-deoxy-D-glucose scanning skeletal muscle

SECONDARY OUTCOMES:
skeletal muscle blood flow | 26 weeks
  measured using PET scanning
insulin signaling pathways in skeletal muscle | 26 weeks
  measured from muscle biopsies taken before and after intervention
insulin sensitivity of bone marrow fat | 26 weeks
  measured using PET images
insulin stimulated intestinal glucose uptake | 26 weeks
  measured using PET images

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Nuutila, MD, PhD, Principal Investigator — Turku University Hospital
Locations (3):
- Finland (3):
  - Turku PET Centre, Turku, Turku
  - Turku university hospital, PET center, Turku, Turku
  - Turku PET Centre (Turku University Hospital), Turku

REFERENCES:
- [Derived] Koffert JP, Mikkola K, Virtanen KA, Andersson AD, Faxius L, Hallsten K, Heglind M, Guiducci L, Pham T, Silvola JMU, Virta J, Eriksson O, Kauhanen SP, Saraste A, Enerback S, Iozzo P, Parkkola R, Gomez MF, Nuutila P. Metformin treatment significantly enhances intestinal glucose uptake in patients with type 2 diabetes: Results from a randomized clinical trial. Diabetes Res Clin Pract. 2017 Sep;131:208-216. doi: 10.1016/j.diabres.2017.07.015. Epub 2017 Jul 20. PMID 28778047